CLINICAL TRIAL: NCT04243291
Title: The Prevalence of Road Crash Involvement and Its Associated Factors Among Medical Doctors in Malaysia : A Cross Sectional Study
Brief Title: The Prevalence of Road Crash Involvement and Its Associated Factors Among Medical Doctors in Malaysia
Status: Completed | Type: Observational
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Aneesa Abdul Rashid, Medical Lecturer and Family Medicine Specialist, Universiti Putra Malaysia
Other Study IDs: 40609; 04-01-18-1972FR (Other Grant/Funding Number: MINISTRY OF EDUCATION)
Record Dates: First submitted 2020-01-16; First posted 2020-01-28 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Traffic Accident
Keywords: risk factor; physician; road accident; prevalence

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study mainly to investigate the prevalence of road crash involvement and its associated factors (fatigue, demographic factors, sleep quality, and mental health status, number of working hours) among medical doctors in Malaysia.

DETAILED DESCRIPTION:
The incidence reports of road crash involvement among medical doctors in Malaysia have steadily increased in frequency by 28%. Despite the gravity of the situation, there is an obvious absence of further information regarding the causes of such occurrence. A deeper look into literature regarding the phenomenon worldwide indicates that the prevalence of road crash involvement among doctors are less reported on, much less the factors associated with it.

hence, investigators constructed a research to investigate the prevalence of road crash involvement and its associated factors (fatigue, demographic factors, sleep quality, and mental health status, number of working hours) among medical doctors in Malaysia.

It is a cross sectional study where the study population consists of Malaysian Medical Association (MMA) members who are fully or partially registered with the Malaysian Medical Council (MMC) and their contacts.

Respondents will be selected via non probability random sampling among MMA registered member list and their network. The sample will be doctors who are partially or fully registered with the Malaysian Medical Council and following the inclusion and exclusion criteria. The participants who are eligible will need to answer via an online survey link.

Inclusion criteria

* Malaysian citizen
* Full or partial registration with MMC
* Work a minimum of six (6) months in public healthcare sector in Malaysia. Doctors who have just been working for less than six months are still adapting to the duties and atmosphere of the hospital, and the responsibilities they hold are also different from those of a senior doctor making them not suitable to include in this study.

Exclusion criteria

* Medical doctors currently on a long leave. As investigators only have a short period of data collection, so investigators will exclude this group of subject.
* Does not self-commute to work

CALCULATED SAMPLE SIZE = 288.

This study will be in collaboration with Malaysian Medical Associations (MMA) on recruiting sample for this research along with other medical NGOs. MMA will help in dissemination of information throughout their website as well as distribute/email the questionnaires to all MMA members and their contacts.

The questionnaire will be created by using Google Form and then saved on Google Drive. Then MMA will share the form to all their members through email. All responses will be saved in the file stored in Google Drive. Once enough sample acquired, the form will be closed and results will be download for data analysis.

Data entry and analysis will be undertaken by using the 'Statistical Package for Social Sciences' (SPSS) programme, Version 22.0. The statistical significance level is taken at the p value <0.05 with 95% of confidence intervals (CI). The continuous variables will be summarised by using means and standard deviation (SD) and predominantly categorised as required and presented as the number (n) and percentage (%). The statistics analysis will utilise the Pearson Chi-square test for obtaining the statistical difference of the categorical variables.

Lastly, logistic regression analysis will be used to describe the strength of association between the outcome and factors of interest, adjusting for covariates or confounders. It also allows one to determine the important factors affecting the outcome and generate the final model for the factors being studied as the predictor for the outcomes.

Study Instrument: Questionnaire/scoring & Pilot study

This study's approval for ethical clearance will be obtained from Medical Research Ethics Committee (MREC), "University Putra Malaysia" (UPM). Informed consent will be obtained from each study participant and it will be stated at the beginning of the questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Malaysian citizen
* Full or partial registration with MMC
* Work a minimum of six (6) months in public healthcare sector in Malaysia. Doctors who have just been working for less than six months are still adapting to the duties and atmosphere of the hospital, and the responsibilities they hold are also different from those of a senior doctor making them not suitable to include in this study.

Exclusion Criteria:

* Medical doctors currently on a long leave. As we only have a short period of data collection, so we will exclude this group of subject.
* Does not self-commute to work

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Malaysian Medical Association (MMA) members who are fully or partially registered with the Malaysian Medical Council (MMC) and their contacts. MMA is the main representative body for all registered medical practitioners in Malaysia. MMA members include senior and junior doctors, private and public, specialists and general practioners, medical officer and house officer.
Sampling Method: Non-Probability Sample
Enrollment: 375 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
The Prevalence of Road Crash Involvement among Medical Doctors | Since joining medical profession ( anywhere from one year up to 20 years )
  Self reported in sociodemographic questionnaire
fatigue among Medical Doctors | Since joining medical profession ( anywhere from one year up to 20 years )
  Checklist Individual Strength Questionnaire (CISQ)

CONTACTS AND LOCATIONS:
Overall Officials: Aneesa Abdul Rashid, Principal Investigator — Universiti Putra Malaysia
Locations (1):
- Universiti Putra Malaysia, Seri Kembangan, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aneesa AR, Suhazeli A, Nur Asyikin M, Munawar S, Nur Asyraf M , Siti Illiana M, et al. Post Call MVA Survey: An 18 Hour Online Survey. In: 17th Islamic Association of Malaysia (IMAM) Annual Scientific Conference (ASC). Penang, Malaysia; 2015.
- [Background] Marcus CL, Loughlin GM. Effect of sleep deprivation on driving safety in housestaff. Sleep. 1996 Dec;19(10):763-6. doi: 10.1093/sleep/19.10.763. PMID 9085483
- [Background] Steele MT, Ma OJ, Watson WA, Thomas HA Jr, Muelleman RL. The occupational risk of motor vehicle collisions for emergency medicine residents. Acad Emerg Med. 1999 Oct;6(10):1050-3. doi: 10.1111/j.1553-2712.1999.tb01191.x. PMID 10530665
- [Background] Veasey S, Rosen R, Barzansky B, Rosen I, Owens J. Sleep loss and fatigue in residency training: a reappraisal. JAMA. 2002 Sep 4;288(9):1116-24. doi: 10.1001/jama.288.9.1116. PMID 12204082
- [Background] Pertubuhan Keselamatan Sosial. Laporan Tahunan Perkeso. 2015.
- [Background] Azhar A. Commuting Accidents : What Does Research Shows ? COMMUTING ACCIDENTS PREVENTION SEMINAR MONASH UNIVERSITY MALAYSIA 9 - 10 DECEMBER 2014. 2014.
- [Background] Barger LK, Cade BE, Ayas NT, Cronin JW, Rosner B, Speizer FE, Czeisler CA; Harvard Work Hours, Health, and Safety Group. Extended work shifts and the risk of motor vehicle crashes among interns. N Engl J Med. 2005 Jan 13;352(2):125-34. doi: 10.1056/NEJMoa041401. PMID 15647575
- [Background] Owens JA. Sleep loss and fatigue in healthcare professionals. J Perinat Neonatal Nurs. 2007 Apr-Jun;21(2):92-100; quiz 101-2. doi: 10.1097/01.JPN.0000270624.64584.9d. PMID 17505227
- [Background] World Health Organization Western Pacific Region. Human Resource s for health country profiles : Malaysia. 2014.
- [Background] Fruchtman Y, Moser AM, Perry ZH. Fatigue in medical residents--lessons to be learned. Med Lav. 2011 Sep-Oct;102(5):455-63. PMID 22022764
- [Derived] Rashid AA, Devaraj NK, Mohd Yusof H, Mustapha F, Wong SV, Ismail AF, Ismail KI, Qureshi AM, Nordin RB. Prevalence and predictors of road crash involvement among medical doctors in Malaysia: a cross-sectional study protocol. BMJ Open. 2020 Jul 2;10(7):e037653. doi: 10.1136/bmjopen-2020-037653. PMID 32616493
- See also: Taylor AH, Dorn L. STRESS, FATIGUE, HEALTH, AND RISK OF ROAD TRAFFIC ACCIDENTS AMONG PROFESSIONAL DRIVERS: The Contribution of Physical Inactivity. Annu Rev Public Health [Internet]. 2006;27(1):371-91 — http://www.annualreviews.org/doi/10.1146/annurev.publhealth.27.021405.102117